CLINICAL TRIAL: NCT06276842
Title: Efficacy of Combining an Inferior Alveolar Nerve Block With a Buccal Infiltration for Mandibular Molars With Irreversible Pulpitis
Brief Title: Efficacy of Combining an Inferior Alveolar Nerve Block With a Buccal Infiltration
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CIMS Dental College (Other)
Responsible Party: Principal Investigator, Ayesha Ahmed, Demonstrator,Operative Dentistry Department, CIMS Dental College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 12345678
Record Dates: First submitted 2023-05-09; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Pulpitis
Keywords: Anesthesia; Inferior Alveolar Nerve; Infiltration
MeSH Terms: conditions — Pulpitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient of Group A given Inferior Alveolar Nerve Block (Experimental): The intervention involved approaching the nerve from the contralateral side of the oral cavity over the contralateral premolars. The needle was inserted into the mandibular tissue along the average boundary of the mandibular ramus within the pterygomandibular space and lateral to the pterygomandibular fold. If bony contact was not achieved within 27-29 mm of needle insertion, the needle was slightly withdrawn and repositioned more distally toward the premolars. After achieving bony contact, the needle was withdrawn by 1-2 mm, aspiration was performed, and then 1.8 ml of anesthetic solution was deposited.
  Interventions: Drug: Inferior Alveolar Nerve Block
- Group B-buccal infiltration-supplementary injection technique to Inferior Alveolar Nerve block (Experimental): The intervention began by penetrating the needle into the buccal mucosa adjacent to the mandibular first molar. After aspiration, 1.8 ml of anesthetic solution (2% lignocaine with 1:100,000 epinephrine) was administered over approximately 2 minutes. Following a 15-minute period post-injection, each patient was asked about the level of numbness in their lip. Patients who did not experience significant lip numbness within this 15-minute timeframe were excluded from the study. For patients who reported positive lip numbness, the affected tooth was isolated using a rubber dam, and a traditional access opening procedure was initiated.
  Interventions: Drug: Buccal Infiltration; Combination Product: Inferior Alveolar Nerve Block and Buccal Infiltration

INTERVENTIONS:
Drug: Inferior Alveolar Nerve Block — Administration of a local anesthetic agent around the inferior alveolar nerve to achieve anesthesia in the mandibular region.
  Arms: Patient of Group A given Inferior Alveolar Nerve Block
Drug: Buccal Infiltration — Administration of a local anesthetic agent into the tissue adjacent to the tooth being treated to achieve localized anesthesia.
  Arms: Group B-buccal infiltration-supplementary injection technique to Inferior Alveolar Nerve block
Combination Product: Inferior Alveolar Nerve Block and Buccal Infiltration — Utilization of both the Inferior Alveolar Nerve Block and Buccal Infiltration techniques simultaneously for anesthesia in the mandibular region.
  Arms: Group B-buccal infiltration-supplementary injection technique to Inferior Alveolar Nerve block

SUMMARY:
OBJECTIVE To compare the effectiveness of using both a combined technique of an Inferior Alveolar Nerve block and buccal infiltration with that achieved by utilizing an Inferior Alveolar Nerve block alone for endodontic treatment of mandibular molars with irreversible pulpitis.

STUDY DESIGN Randomized clinical trial PLACE AND DURATION OF STUDY Operative Dentistry Department of Armed Forces Institute of Dentistry Rawalpindi, from 1st April 2020 to 31st September 2020.

MATERIAL AND METHODS A total of 120 patients were enrolled in the study. Sixty patients of group A received conventional Inferior Alveolar Nerve block and sixty patients of Group B received buccal infiltration along with conventional Inferior Alveolar Nerve block.

DETAILED DESCRIPTION:
Patients of Group A received Inferior Alveolar Nerve block anesthesia. For this block, nerve was approached from the contra-lateral side of the oral cavity over the contralateral premolars. Needle penetrated into the mandibular tissue on the average boundary of the mandibular ramus inside the pterygomandibular space and lateral to pterygomandibular fold, it advanced until bony surface was contacted. In the event that bony contact wasn't made inside 27-29 mm of needle infiltration, needle was pulled back somewhat, moved the needle further distally toward premolars. The needle was withdrew 1-2 mm after making bony contact, aspiration was performed, followed by 1.8 ml deposition of anesthetic solution.

Patients of Group B received buccal infiltration as supplementary injection technique to conventional Inferior Alveolar Nerve block, buccal infiltration was carried out. The needle was penetrated in buccal mucosa adjacent to mandibular 1st molar. After aspiration, 1.8ml of anesthetic solution was dumped in approximate time of 2 minutes using 2% lignocaine with 1:100,000 epinephrine. Following time period of 15 minutes of injection, every patient was inquired about his/her lip numbness. Patients who did not experience significant lip numbness within 15 minutes after the block was administered were excluded from the investigation and was considered ineffective. In case of positive lip numbness patient concerned teeth was isolated using rubber dam and a traditional access opening was started. Patient was told to lift hand if any pain will occur while doing procedure. The patient was requested to mark pain on visual analogue scale (VAS) after completion of treatment. Absence of pain was indicated if patient scored his/her pain ≤ 3 on VAS.

ELIGIBILITY:
Inclusion Criteria:

* Mandibular molars with irreversible pulpitis (confirmed by positive response to EPT)
* Patient age between 18 to 45 years
* No medication taken 24 hours before treatment
* Both male and female patients

Exclusion Criteria:

* Patients on analgesics or anti-inflammatory drugs
* Medically compromised patients
* Teeth with immature apices
* Retreatment cases
* Patients allergic to lignocaine
* Teeth with root resorption
* Teeth with necrotic pulp
* Apical abscess
* Pregnancy

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Comparison of Anesthesia Effectiveness Between Combined Technique (Inferior Alveolar Nerve Block and Buccal Infiltration) and Inferior Alveolar Nerve Block Alone | 6 months
  This investigation aims to assess the effectiveness of a combined technique involving an Inferior Alveolar Nerve block and buccal infiltration in providing supplementary anesthesia for the treatment of symptomatic irreversible pulpitis in the local population. The study will utilize quantitative measures to evaluate the number of participants experiencing successful anesthesia, measured by specific parameters such as pain relief scores. If demonstrated to be more effective than traditional methods, this technique may be recommended for routine clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Dil Rasheed, BDS,FCPS, Study Director — CMH Multan Institute of Medical Sciences
Locations (1):
- Dr Ayesha Ahmed, Multan, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dougall A, Apperley O, Smith G, Madden L, Parkinson L, Daly B. Safety of buccal infiltration local anaesthesia for dental procedures. Haemophilia. 2019 Mar;25(2):270-275. doi: 10.1111/hae.13695. Epub 2019 Feb 28. PMID 30817070
- [Background] Abazarpoor R, Parirokh M, Nakhaee N, Abbott PV. A Comparison of Different Volumes of Articaine for Inferior Alveolar Nerve Block for Molar Teeth with Symptomatic Irreversible Pulpitis. J Endod. 2015 Sep;41(9):1408-11. doi: 10.1016/j.joen.2015.05.015. Epub 2015 Jul 3. PMID 26149210
- [Background] Lin S, Wigler R, Huber R, Kaufman AY. Anaesthetic efficacy of intraligamentary injection techniques on mandibular molars diagnosed with asymptomatic irreversible pulpitis: A retrospective study. Aust Endod J. 2017 Apr;43(1):34-37. doi: 10.1111/aej.12169. Epub 2016 Aug 25. PMID 27558847
- [Result] Chopra R, Marwaha M, Bansal K, Mittal M. Evaluation of Buccal Infiltration with Articaine and Inferior Alveolar Nerve Block with Lignocaine for Pulp Therapy in Mandibular Primary Molars. J Clin Pediatr Dent. 2016;40(4):301-5. doi: 10.17796/1053-4628-40.4.301. PMID 27471808